CLINICAL TRIAL: NCT05641298
Title: A Phase 2, Randomized, DB, Placebo-controlled Study to Determine the Efficacy, Safety and PK Profile of ARV-1801 in Combination With Optimized Background Therapy for the Treatment of Pulmonary Exacerbations in Patients With Cystic Fibrosis
Brief Title: Study to Determine the Efficacy&Safety of ARV-1801(ACG-701) for the Treatment of Cystic Fibrosis Pulmonary Exacerbations
Acronym: REPRIEVE
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Corporate finances
Sponsor: Aceragen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACG-701-101
Record Dates: First submitted 2022-11-29; First posted 2022-12-07 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-02

CONDITIONS: Cystic Fibrosis; Cystic Fibrosis Pulmonary Exacerbation
Keywords: Pulmonary Exacerbation; Antibiotic
MeSH Terms: conditions — Cystic Fibrosis | interventions — Fusidic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ARV-1801(ACG-701) Active Group (Active Comparator): ARV-1801(ACG-701) tablets by mouth twice a day for 14 days
  Interventions: Drug: Sodium Fusidate
- Placebo Group (Placebo Comparator): Placebo tablets by mouth twice a day for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Fusidate — Tablets
  Other Names: ACG-701; ARV-1801
  Arms: ARV-1801(ACG-701) Active Group
Drug: Placebo — Tablets
  Arms: Placebo Group

SUMMARY:
This study will evaluate the efficacy and safety of an oral ARV-1801(ACG-701) plus optimized background therapy (OBT) compared to oral placebo plus OBT, each administered for 14 days, in the treatment of participants with Cystic Fibrosis-related pulmonary exacerbations (PEx).

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, multicenter study designed to evaluate the efficacy and safety of an oral ARV-1801/ACG-701 plus OBT compared to oral placebo plus OBT, each administered for 14 days, in the treatment of participants with CF-related PEx.

Participants who provide informed consent (plus informed assent, if applicable) and meet all study eligibility criteria will be enrolled in the study and randomized via an interactive response technology (IRT) in a 1:1 ratio to receive ARV-1801/ACG-701 or placebo in addition to OBT for 14 days. A participant may be hospitalized (inpatient) or treated as an outpatient. If admitted to the hospital for initial treatment, the participant may be discharged at the Investigator's discretion to complete study therapy as an outpatient. The target study population will comprise 80 participants.

The duration of participation in the study for an individual participant will be approximately 28 days and will involve up to 5 clinic visits as well as the requirement to complete an electronic symptom questionnaire every day for the duration of the study. Participation will include a Screening period of up to 24 hours prior to the first dose of study drug (Day 1), a 14 day treatment course of study drug, a Day 7 visit (±1 day), an end of treatment (EOT) visit (day of last dose of study drug +3 days), and end of study (EOS) visit on Day 28 (+3 days).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females of 12 years of age and older
2. Participants must have a confirmed diagnosis of Cystic Fibrosis with a diagnosis of an acute pulmonary exacerbation as defined as:

   1. Deterioration in 3 or more of the following symptoms for at least 48 hrs (cough, sputum volume and/or consistency, sputum purulence, breathlessness and/or exercise tolerance, fatigue and/or malaise, or hemoptysis) And
   2. a clinician determines that a change in CF treatment is required
3. Participants must have a CFRSD-CRISS score of >/= 35
4. Participants must have a moderate or Severe Patient Global Impression of Severity
5. Participants must have a negative pregnancy test and agree to use a highly effective method of contraception during the study and 30 days after last dose
6. Participants must agree not to smoke during any part of the clinical trial
7. Participants must voluntarily sign the informed consent for the study

Exclusion Criteria:

1. Participants cannot have any changes in any antimicrobial, bronchodilator, anti-inflammatory, CFTR modulator or corticosteroid medications from 28 - 3 days prior to the Screening visit.
2. Participants cannot be receiving treatment for non-tuberculosis mycobacteria and/or Aspergillus infection.
3. History of hypersensitivity or allergic reaction to sodium fusidate, fusidic acid (Fucidin®) or its excipients.
4. Abnormal laboratory findings or other findings or medical history at Screening that, in the Investigator's opinion, would compromise the safety of the participant or the quality of the study data.
5. The use of an investigational drug or device (ie, a drug or device without the FDA approved indication) within 30 days prior to the Screening visit
6. Known severe renal impairment, as indicated by estimated creatinine clearance (CrCl) <30 mL/min (by Cockcroft-Gault calculation).
7. Evidence of significant liver disease: ALT >3×ULN, or direct bilirubin >ULN, or total bilirubin >1.5 mg/dL; known cirrhosis with decompensation (ie, Child-Pugh Class B or C disease).
8. Known hepatitis C virus (HCV) or infection and currently receiving HCV-specific antiviral therapy. HCV infection alone, and in the absence of decompensated liver disease, is not exclusionary.
9. Neutropenia (absolute neutrophil count <500/µL); thrombocytopenia (<60,000 platelets/mm3).
10. Known human immunodeficiency virus (HIV) infection and currently receiving antiretroviral therapy, or current CD4 count ≤200 cells/mm3 (documented within 3 months prior to enrollment); if CD4 count is unknown, participant may not enroll.
11. Changes to or initiation of immunosuppressant agents (ie, prednisone [≥15mg/day], cyclosporine, tumor necrosis factor alpha [TNFα] antagonist) within 30 days of study medication administration through the EOS visit.
12. Malignancy requiring ongoing cytotoxic chemotherapy or radiation therapy.
13. Requires concomitant treatment with (washout period prior to randomization allowed):

    * OATP1B1 and OATP1B3 substrates (eg, HMG-CoA reductase inhibitors [statins])
    * CYP2C8 substrates, namely glitazones (eg, repaglinide)
    * CYP3A4 inducers (eg, dexamethasone, phenytoin, carbamazepine, rifampin, phenobarbital, nafcillin)
    * Moderate/strong CYP3A4 inhibitors (eg, azole antifungals, erythromycin, clarithromycin)
    * P-gp substrates with narrow therapeutic windows (eg, digoxin and colchicine)
14. Prior treatment with a CYP3A4 inducer (such as lumacaftor, dexamethasone, phenytoin, carbamazepine, rifampin, phenobarbital and nafcillin) within 7 days prior to enrollment.
15. Dietary use of large amounts of grapefruit juice and/or Seville oranges or other products containing these fruits (eg, grapefruit juice or marmalade) during the study.
16. Participant requiring warfarin therapy.
17. Seizure disorder requiring current therapy with an anticonvulsant.
18. Female participant who is pregnant or lactating.
19. History of /current chronic alcohol consumption and/or drug abuse (including cannabis use).
20. Any study personnel or their immediate dependents, family, or household members.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Desirability in outcome ranking (DOOR) | Day 7
  To demonstrate that the addition of oral ARV-1801(ACG-701) to OBT is superior to placebo plus OBT based on DOOR in cystic fibrosis pulmonary exacerbations.

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - University of Florida, Gainesville, Florida
  - Central Florida Pulmonary Group, Orlando, Florida
  - Nemours Children's Health - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Cystic Fibrosis Center of Chicago, Chicago, Illinois
  - Cystic Fibrosis Center of Chicago, Northfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University Of Louisville, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Michigan Medicine, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - UNMC-Nebraska CF Pediatric Center, Omaha, Nebraska
  - Gunnar H. Esiason Adult Cystic Fibrosis Center, Morristown, New Jersey
  - New York Medical College, Hawthorne, New York
  - University of Rochester Medical Center Strong Memorial, Rochester, New York
  - Rainbow Babies and Children's Hospital/Cleveland Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Cook Children's Health Care System, Fort Worth, Texas
  - The University of Health Science Center at Tyler, Tyler, Texas
  - Providence Medical Research Center, Spokane, Washington